CLINICAL TRIAL: NCT02075710
Title: Lipogenesis, Lipoprotein Flux, and CVD Risk: Role of Meal Composition and Frequency
Brief Title: Dietary Treatment Study of Fat Synthesis and Risk of Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: Touro University, California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: Nibble99
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Overweight and Obesity
Keywords: Diet; Sugar; Cardiovascular; Lipid
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- High sugar/meal feed (Experimental): Diet high in simple sugar fed as two large meals daily
  Interventions: Other: High sugar/meal feed; Other: High sugar/nibble
- High sugar/nibble (Experimental): Diet high in simple sugar fed as 8 small meals daily
  Interventions: Other: High sugar/meal feed; Other: High sugar/nibble
- High fat/meal feed (Experimental): Diet high in fat fed as two large meals daily
  Interventions: Other: High fat/meal feed; Other: High fat/nibble
- High fat/nibble (Experimental): Diet high in fat fed as 8 small meals daily
  Interventions: Other: High fat/nibble
- High sugar/3 meals a day (Experimental): Diet high in simple sugar fed as 3 meals a day
  Interventions: Other: High sugar/ 3 meals a day; Other: High fat/ 3 meals a day
- High fat/ 3 meals a day (Experimental): Diet high in fat fed as 3 meals a day
  Interventions: Other: High sugar/ 3 meals a day; Other: High fat/ 3 meals a day

INTERVENTIONS:
Other: High sugar/meal feed — Weight-maintaining diet relatively high in sugar fed as two large meals daily
  Arms: High sugar/meal feed; High sugar/nibble
Other: High sugar/nibble — Weight-maintaining diet relatively high in sugar fed as 8 meals daily
  Arms: High sugar/meal feed; High sugar/nibble
Other: High fat/meal feed — Weight-maintaining diet relatively high in fat fed as two large meals daily
  Arms: High fat/meal feed
Other: High fat/nibble — Weight-maintaining diet relatively high in fat fed as 8 small meals daily
  Arms: High fat/meal feed; High fat/nibble
Other: High sugar/ 3 meals a day — Weight-maintaining diet relatively high in sugar fed as 3 meals daily
  Arms: High fat/ 3 meals a day; High sugar/3 meals a day
Other: High fat/ 3 meals a day — Weight-maintaining diet relatively high in fat fed as 3 meals daily
  Arms: High fat/ 3 meals a day; High sugar/3 meals a day

SUMMARY:
The purpose of this study is to find out how the amount of fat or sugar in a person's diet, or the number of meals eaten each day, affect the amount of fat that people's bodies make, the types of fats in the bloodstream, and how much fat is stored in the liver. The study is funded by the National Institutes of Health.

DETAILED DESCRIPTION:
The study consists of two 10-day feeding periods that are separated by approximately two weeks. During each feeding period all food and beverages to be consumed will be provided by the study.

In Study 1, participants will be randomly assigned to receive one of two diets. Both diets are designed to maintain weight at a constant level. The diets are balanced nutritionally and have the same amount of protein. One diet has higher amounts of sugar, while the other has higher amounts of fat. For one 10-day period, the diet will be fed as two large meals ('meal-feeding'). For the other 10-day period, the identical diet will be fed as 8 small meals ('nibbling'). Half of the participants will meal-feed first, while the other half will 'nibble' first. The order of nibbling or meal feeding will be determined randomly.

In Study 2, the number of meals eaten per day will remain fixed at three (no nibbling or meal feeding). Participants will receive both the diet higher in sugar and the diet higher in fat. However, they will be randomly assigned to start one followed by the other for each 10-day feeding period.

At the end of each 10-day feeding period, participants will spend two nights in a research ward (Clinical Research Center) to undergo testing.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese men and women
* ages 20-65 years

Exclusion Criteria:

* pregnancy or lactation within the past six months
* type 1 or 2 diabetes mellitus]
* AST and ALT above upper limit of normal (ULN)
* fasting triglyceride or total cholesterol levels >ULN
* Hgb below the lower of limit of normal
* positive HIV antibody test or hepatitis serologies
* use of any antidiabetic medications or lipid-lowering drugs
* history of surgery for obesity
* change in body weight >5% within preceding 6 months (self report)
* claustrophobia, presence of metal implants
* weight over 350 lbs

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-07; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Effect of meal composition on fractional de novo lipogenesis (fatty acid synthesis) | After 10-day dietary period
  Differences between high carbohydrate and high fat diets on postprandial de novo lipogenesis
  De novo lipogenesis will be measured using stable (not radioactive) isotopes given intravenously and orally during feeding.

SECONDARY OUTCOMES:
Effect of meal frequency on fractional de novo lipogenesis (fatty acid synthesis) | After 10-day dietary period
  Differences between consuming the same diet as eight small meals per day or two larger meals per day on postprandial de novo lipogenesis.
  Please see description of measurement of de novo lipogenesis under aim 1.

OTHER OUTCOMES:
Liver fat content | After 10-day dietary period
  Effects of diet composition or meal frequency on fat stored in the liver.
  Liver fat content will be measured non-invasively using magnetic resonance spectroscopy.
Lipids and lipoproteins in the blood | After 10-day dietary intervention period
  Effects of diet composition or meal frequency on the types of fats in the bloodstream that might affect risk of heart disease.
  The types of fats in the bloodstream will be measured in blood samples collected while the participant is fasting and also during the stable isotope/feeding study of de novo lipogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Mulligan, PhD, Principal Investigator — University of California, San Francisco; Jean-Marc Schwarz, PhD, Principal Investigator — Touro University, California
Locations (1):
- University of California, San Franciso, San Francisco General Hospital, San Francisco, California, United States